CLINICAL TRIAL: NCT03089268
Title: Molecular and Histological Characteristics of Serrated Lesions of the Colon: Development of an Individual Risk Profile Applicable to Population-based Colorectal Cancer Screening Programs
Brief Title: Molecular and Histological Characteristics of Serrated Lesions of the Colon
Acronym: SERRACOLON
Status: Active, not recruiting | Type: Observational
Sponsor: Hospital Universitario La Fe (Other)
Responsible Party: Principal Investigator, Marco Bustamante-Balén, Gastrointestinal Endoscopy Consultant, Hospital Universitario La Fe
Other Study IDs: PSC-01A
Record Dates: First submitted 2017-03-20; First posted 2017-03-24 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Colonic Neoplasms; Colorectal Cancer; Sessile Serrated Adenoma; Polyp of Colon
Keywords: sessile serrated polyp; prevalence; colorectal cancer; molecular biology
MeSH Terms: conditions — Colonic Neoplasms; Colorectal Neoplasms; Colonic Polyps | interventions — Colonoscopy; Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — colonic polyp or colorectal cancer samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Individuals scheduled for colonoscopy at Hospital Universitari i Politècnic La Fe, participating in the Valencian CRC screening program, will be recruited.
  Polypectomy or biopsy will be performed if necessary (following current guidelines).
  Specific molecular analysis of serrated lesions and CRC will be carried out.
  Interventions: Procedure: Colonoscopy; Procedure: Polypectomy or biopsy; Genetic: Molecular analysis

INTERVENTIONS:
Procedure: Colonoscopy — A colonoscopy will be performed to all individuals.
Procedure: Polypectomy or biopsy — All lesions will be removed or biopsied during the procedure
Genetic: Molecular analysis — Molecular analysis will be performed in all colorectal cancers and in those polyps diagnosed with "serrated lesion"

SUMMARY:
Different subtypes of serrated lesions have been recently described. Among them, both sessile serrated polyp/adenoma (SSP/A) and traditional serrated adenoma (TSA) could have malignant potential through the serrated pathway or CIMP. These lesions, as a potential source of interval cancer, should also be considered in colorectal cancer (CRC) population-based screening programs. It is believed that this new described pathway could be responsible for up to 30% of all CRC.

Unlike the traditional adenoma, serrated lesions are difficult to diagnose because of their particular endoscopic appearance and their still unclear histological criteria. Furthermore, they have specific molecular changes and, through them, they could evolve into CRC faster than the adenoma. The real prevalence of the serrated lesions and their specific risk for developing new synchronous/metachronous lesions, or even malignancy, remains unknown. For all these reasons, we don't know if these patients could constitute a different CRC-risk group and if specific recommendations are needed during their follow-up.

This is a prospective longitudinal study developed within the framework of the CRC-screening program in the Valencian Community (Spain). We expect to include a total of 700 individuals who will be followed during 10 years.

In our study, we will collect epidemiologic variables related to the patient, variables related to all the polyps, and mutational (BRAF, KRAS, MSI), and CpG-island methylation status of serrated lesions. Strict endoscopic and histological criteria will be applied for the diagnosis of serrated lesions. All lesions detected at the index colonoscopy and during follow-up will be evaluated.

The purpose of this study is to correlate epidemiologic data, histological characteristics and the molecular profile of the serrated lesions with findings during follow-up, in order to define stratified groups according to their risk of developing new lesions or CRC in the future.

DETAILED DESCRIPTION:
BACKGROUND Colorectal cancer (CRC) is, by its frequency and consequences, a relevant public health problem that has led to the implementation of population screening programs in many countries. The purpose of these programs is to reduce the incidence and mortality of CRC by early diagnosis of the disease, in the so-called pre-symptomatic phase. That is, to identify and remove all precursor lesions, essentially colon adenomas.

However, there is increasing evidence that these programs are not fully effective in preventing CRC. Cancers that appear before the next scheduled endoscopic control, called interval cancer (IC), occur in up to 2.5 / 1000 patients / year of observation, and the cumulative probability of developing a CRC within the first 5 years after an adenoma removal could be up to 2%. Recent studies suggest that the cause of more than 50% of ICs is the failure detecting premalignant lesions in the colon, either due to a poor colon preparation, technical deficiencies in the performance of colonoscopy or the characteristics of the lesions that make them barely visible.

A possible origin of the ICs could be the serrated polyp (SP). This is actually not a single lesion, but a heterogeneous group of lesions, different from the conventional adenoma, and characterized by the serration of the crypts in the histology. Serrated lesions, especially some subgroups, have macroscopic features that make them particularly difficult to detect in conventional colonoscopy: indistinct borders, cloud-like appearance, often covered by a mucous cap and interruption of the underlying mucosal vascular pattern. But the true diagnosis of serrated lesions is made by morphological criteria with the microscopic examination of the sample obtained by biopsy. Although all lesions that showed these features were initially identified as hyperplastic polyps (HP), in the last decade three subtypes of serrated lesions with different clinical implications have been described [HP, sessile serrated polyp/adenoma (SSA/P) and traditional serrated adenoma (TSA)]. However, the histological criteria are not yet fully clarified, and there is confusion in the terms to be used. Therefore, the agreement among pathologists is generally poor.

As a consequence, many serrated lesions are misdiagnosed and incorrectly classified. This has clinical relevance since some of them have malignant capacity. Both SSA/P and TSA can evolve to CRC through the so-called serrated pathway or cytosine-phosphate-guanosine (CpG) island methylator phenotype (CIMP), which could be responsible for up to 30% of all CRC. In this pathway, an aberrant hypermethylation of the genome is produced, which leads to transcriptional silencing and inhibition of expression in some genes promoter regions (epigenetic modification). CRCs that arise from a SP are not homogeneous and may have different molecular and histological characteristics depending on whether the origin mutation in the precursor lesion occurs in BRAF or Kirsten rat sarcoma (KRAS) gene, which leads to the development of SSA/P or TSA. And depending on if a mutL homolog 1 (MLH1) gene methylation is produced thereafter, a unstable (MSI) or stable (MSS) CRC will develop. The presence of a high CIMP rate also depends on the initial mutation. Therefore, serrated lesions could originate MSI/CIMP-H CRC (11%), MSS/CIMP-H CCR (4%) and MSS/CIMP-L CRC (15%). It is thought that some of the ICs may be directly related to the SP because they share morphological and molecular characteristics. The evolution from SSP/SSA to invasive carcinoma has been described to occur in only eight months.

This theoretical risk of developing advanced premalignant lesions and IC and its clinical significance has not been clearly shown in clinical practice because data on the prevalence of serrated lesions are limited and there is also a lack of longitudinal follow-up studies in patients with serrated lesions. The prevalence described is very variable and ranges from 0.6% to 13%, depending on the study, and the data are even scarcer in fecal occult blood test (FOBT) -based screening population. The presence of serrated lesions (other than HP) has been associated with the development of advanced synchronous adenomas in the colon, but also with advanced metachronous lesions during follow-up. This situation could place these patients in a special risk group. Patients with large SP may have a similar risk to develop a future CRC to those patients with advanced adenomas. Most Scientific Societies recommend endoscopic follow-up of serrated lesions, but the evidence is weak and specific intervals are proposed based only on expert recommendations.

In summary, there are still many unresolved questions about serrated polyps and their importance in CRC screening programs. Their prevalence on CRC screening population is not fully clarified because of the lack of prospective trials and the difficulty in diagnosis and histological classification. Their malignant potential is not clarified either because of the uncertainty about the prevalence of dysplasia in serrated lesions, and the lack of well-designed longitudinal studies for the detection of metachronic lesions. The current criteria for classifying these lesions seem weak to define the CRC risk for a specific patient, thus the proposed follow-up intervals are not based on strong scientific evidence. A thorough study of serrated lesions relating their molecular and histological characteristics with lesions found on colonoscopic follow-up could establish a new molecular classification aimed to design a patient-oriented follow-up strategy.

HYPOTHESIS The correlation of epidemiological data of the patient, histological characteristics and molecular alterations of SP of the colon, along with findings in the endoscopic follow-up, would allow to identify stratified groups of patients according to their risk of developing advanced lesions and CRC in the future.

OBJECTIVE

* To deepen the knowledge of histology and genetic alterations of SP and thereby try to establish a molecular classification that may serve as a basis for new endoscopic follow-up guidelines. These recommendations would be more reliable and adjusted to the patient's individual risk profile.
* To establish the prevalence of serrated lesions, especially SSP/SSA and SSP with dysplasia, in the FOBT positive CRC screening population.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing a colonoscopy after a positive FOBT

Exclusion Criteria:

* Previous diagnose of inflammatory bowel disease
* Previous colon surgery
* Hereditary CRC syndrome
* Coagulation disorders
* Refusal of the individual to participate and sign informed consent

Ages: 50 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All individuals undergoing a colonoscopy after a positive FOBT result within the framework of the CRC-screening program in the Hospital Universitari i Politècnic La Fe (Valencia) in the Valencian Community (Spain).
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Risk of developing metachronous advanced lesions or cancers | 2017-2027
  To assess the risk of developing metachronous advanced lesions or cancers in FOBT screening population

SECONDARY OUTCOMES:
Genetic defects of colorectal cancer and serrated lesions | 15/04/17- 15/04/18
  Analysis of molecular changes in colorectal cancer and serrated lesions in FOBT screening population
Prevalence of serrated lesions in FOBT screening population | 15/04/17- 15/04/18
  To assess the prevalence of serrated lesions in FOBT screening population

CONTACTS AND LOCATIONS:
Overall Officials: Marco Bustamante, M.D.;Ph.D., Principal Investigator — Hospital Universitari i Politècnic La Fe - Instituto de Investigación Sanitaria
Locations (1):
- Hospital Universitari i Politècnic La Fe, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided